CLINICAL TRIAL: NCT06705595
Title: The Effect of Two Different Local Anesthetic Techniques on Hemodynamic Response and Postoperative Sore Throat in Patients Intubated with Double-Lumen Tubes: a Randomized Controlled Study
Brief Title: The Effect of Local Anesthetic Techniques on Hemodynamic Response and Postoperative Sore Throat in Double-Lumen Tubes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: V.K.V. American Hospital, Istanbul (Other)
Responsible Party: Principal Investigator, Murat Tümer, MD, Anesthesiologist, V.K.V. American Hospital, Istanbul
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: LA&Double-LumenTubes
Record Dates: First submitted 2024-11-14; First posted 2024-11-26 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Anesthesia, Local; Intubation, Intratracheal; Double-lumen Tube; Sore Throat; Lidocaine Spray
Keywords: Double-lumen tube; Lidocaine; Sore throat; Lidocaine spray
MeSH Terms: conditions — Pharyngitis | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Statisticians:
  The statisticians analyzing the data will remain blinded to the group assignments during the initial stages of analysis to avoid any bias in the interpretation of the results. Unblinding will occur only after the data is fully collected and the analysis plan is in place.
  Data Collection Staff:
  The staff collecting data in the operating room, recovery room, and patient wards (e.g., monitoring vital signs and postoperative complications) will be blinded to the specific treatment group of the patient. This minimizes any potential bias during the collection of clinical data.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group T (Inhaled Lidocaine) (Experimental): Participants will receive 2 ml of 10% lidocaine via a Tracheo-Spray device before anesthesia induction.
  Interventions: Drug: Tracheo-Spray
- Group X (Lidocaine Applied to the Double-Lumen Tube): (Experimental): Participants will receive 10% lidocaine sprayed directly onto the distal surface and cuffs of the double-lumen tube.
  Interventions: Drug: Lidocaine Spray on DLT
- Group C (Control) (Sham Comparator): Participants will receive 1 ml of 0.9% saline as a placebo.
  Interventions: Drug: Saline (Placebo)

INTERVENTIONS:
Drug: Tracheo-Spray — Participants will receive 2 ml of 10% lidocaine delivered via a Tracheo-Spray device to the tracheal mucosa before anesthesia induction.
  Arms: Group T (Inhaled Lidocaine)
Drug: Lidocaine Spray on DLT — Before intubation, participants will receive 10% lidocaine spray applied to the distal surface and cuffs of the double-lumen tube (DLT).
  Arms: Group X (Lidocaine Applied to the Double-Lumen Tube):
Drug: Saline (Placebo) — Before intubation, participants will receive 1 ml of 0.9% saline applied to the distal surface and cuffs of the double-lumen tube (DLT).
  Arms: Group C (Control)

SUMMARY:
This clinical trial aims to determine if different local anesthetic application techniques can reduce postoperative sore throat (POST) and manage hemodynamic responses in adult patients undergoing elective thoracic surgery with double-lumen intubation. The main questions it aims to answer are:

* Does inhaled lidocaine or lidocaine applied to the double-lumen tube reduce the incidence and severity of POST?
* How do these anesthetic techniques impact hemodynamic stability during surgery?

Researchers will compare three groups-those receiving inhaled lidocaine, lidocaine applied to the tube, and a saline control group-to see if these methods differ in effectiveness.

Participants will:

* Undergo standard preoperative assessment and provide informed consent
* Be randomly assigned to receive either inhaled lidocaine, lidocaine applied to the tube, or saline
* Have sore throat scores and hemodynamic data recorded at specific intervals after surgery

DETAILED DESCRIPTION:
This clinical trial is designed to evaluate the effects of two local anesthetic techniques on postoperative sore throat (POST) incidence and hemodynamic responses in patients undergoing elective thoracic surgery with double-lumen tube (DLT) intubation. POST is a common and undesirable outcome following general anesthesia with endotracheal intubation, particularly with DLTs due to their size and dual cuffs, which can increase mucosal irritation. Addressing POST effectively could significantly improve patient comfort, satisfaction, and overall quality of postoperative care.

**Study Protocol Overview:**

Patients meeting eligibility criteria (aged over 18, ASA I-III) will be recruited from Health Sciences University Kartal City Hospital and randomly assigned to one of three groups:

1. Group T (Inhaled Lidocaine): Participants will receive 2 ml of 10% lidocaine inhaled via a Tracheo-Spray device before anesthesia induction. This method is expected to coat the mucosal surfaces of the airway, potentially reducing friction and inflammation.
2. Group X (Lidocaine Applied to Tube): Participants will have 10% lidocaine sprayed directly on the distal surface and cuffs of the DLT. This technique aims to provide direct anesthetic coverage on the tube surface, potentially reducing mucosal damage from intubation.
3. Group C (Control): Participants will receive 1 ml of 0.9% saline spray as a placebo.

Data Collection:

The primary outcome measure will be the severity of POST, assessed at 2, 6, 12, and 24 hours postoperatively using a throat pain score (0 to 5 scale). Secondary measures will include hemodynamic parameters (heart rate, systolic and diastolic blood pressures) documented before and after lidocaine application, as well as the incidence of postoperative complications such as hypotension, hypoxemia, hypercapnia, nausea, vomiting, and emergence agitation. Trained investigators will collect data in the operating room, recovery room, and patient wards.

Statistical Analysis:

Data will be analyzed using descriptive and inferential statistics. The Kolmogorov-Smirnov test will assess the normality of data distribution. One-way ANOVA and Bonferroni or Tamhane post-hoc tests will be used for normally distributed variables. For non-parametric variables, the Kruskal-Wallis test and Mann-Whitney U test will be applied. Pearson's chi-square or Fisher's exact test will be used to evaluate qualitative variables, with significance set at p < 0.05.

By comparing different application methods, this study aims to determine an effective approach for reducing POST, which could provide guidance for anesthetic practices in thoracic surgery involving DLTs.

ELIGIBILITY:
Inclusion Criteria:

* Aged over 18 years
* ASA (American Society of Anesthesiologists) scores of 1-3
* Elective thoracic surgery patients

Exclusion Criteria:

* Patients with ASA scores of 4 or above
* Do not consent to participate
* individuals with mental disorders
* patients under 18 years of age
* surgeries exceeding two hours
* those with known allergies to local anesthetic

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-11-06 (Actual); Primary Completion 2024-12-06 (Actual); Study Completion 2024-12-12 (Actual)

PRIMARY OUTCOMES:
Postoperative Sore Throat (POST) | 2, 6, 12, and 24 hours after surgery
  The severity of POST will be assessed at 2, 6, 12, and 24 hours after surgery using a throat pain score, ranging from 0 (no pain) to 5 (worst imaginable pain).

SECONDARY OUTCOMES:
Intraperative Hemodynamic Responses | Basal measurements and 5 minutes after intubation.
  Hypotension: Defined as a decrease of more than 20% in systolic blood pressure from baseline or < 80 mmHg.
  Hypertension: Defined as an increase of more than 20% in systolic blood pressure from baseline or > 120 mmHg.

OTHER OUTCOMES:
Postoperative Complications: | Postoperative 2. 6. 12. and 24. hours
  Hypotension: Defined as a decrease of more than 20% in systolic blood pressure from baseline or < 80 mmHg.
  Nausea and Vomiting: Incidence and severity of nausea and vomiting after surgery.
  Hypoxemia: Defined as SpO2 < 90% or PaO2 < 60 mmHg. Hypercapnia: Defined as PaCO2 > 45 mmHg. Emergence Agitation: The presence and severity of agitation during emergence from anesthesia.

CONTACTS AND LOCATIONS:
Locations (1):
- Health Sciences University Kartal City Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The data that will be shared includes the following: Demographic Information, Postoperative Sore Throat (POST) Scores, Hemodynamic Data, and Intraoperative Complications.
  All shared data will be de-identified to protect participant confidentiality, and access will be granted only to researchers who meet the necessary criteria and ethical standards for data use.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The start date for IPD sharing will be after the completion of the study and the publication of the main study results, approximately June 2025.
  End Date for IPD Sharing:
  IPD will be available for sharing for a period of 5 years following the publication of the study results, until June 2030.
  During this period, researchers who meet the criteria for access will be able to request the de-identified data for secondary analyses.

REFERENCES:
- [Background] Chandler M. Tracheal intubation and sore throat: a mechanical explanation. Anaesthesia. 2002 Feb;57(2):155-61. doi: 10.1046/j.1365-2044.2002.02329.x. PMID 11871952
- [Background] Tanaka Y, Nakayama T, Nishimori M, Tsujimura Y, Kawaguchi M, Sato Y. Lidocaine for preventing postoperative sore throat. Cochrane Database Syst Rev. 2015 Jul 14;2015(7):CD004081. doi: 10.1002/14651858.CD004081.pub3. PMID 26171894
- [Background] El-Boghdadly K, Bailey CR, Wiles MD. Postoperative sore throat: a systematic review. Anaesthesia. 2016 Jun;71(6):706-17. doi: 10.1111/anae.13438. Epub 2016 Mar 28. PMID 27158989